CLINICAL TRIAL: NCT04440306
Title: "Tailored" Bilio-Pancreatic Limb Length and Weight Loss After One Anastomosis Gastric Bypass [" Mini-Gastric Bypass Original Technique"]
Brief Title: "Tailored" Bilio-Pancreatic Limb Length and Weight Loss After Mini-Gastric Bypass
Acronym: BplVsWtLoss
Status: Completed | Type: Observational
Sponsor: Kular Hospital (Other)
Responsible Party: Principal Investigator, Dr. Robert Rutledge, Research Director, Kular Hospital
Other Study IDs: BPLL-vs-WtLoss
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Obesity, Morbid; Weight Loss; Bariatric Surgery Candidate; Power
Keywords: Mini-Gastric Bypass; Bilio-Pancreatic Limb Length; Weight loss; One Anastomosis Gastric Bypass
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mini-Gastric Bypass - Original Technique — Mini-Gastric Bypass - Original Technique is widely used form of bariatric surgery and includes a tailored BPLL
  Other Names: Tailored Bilio-Pancreatic Limb Length

SUMMARY:
Retrospective review of prospectively collected blinded patient data. To Address simple question:

In cases of Mini-Gastric Bypass performed using the Original Technique what (if any) is the relation between the Bilio-pancreatic limb length (BPLL) and the patient weight loss at 10 years following operation.

DETAILED DESCRIPTION:
Methods:

The investigators performed a review of a prospectively collected database system of patients undergoing tailored MGB-OT at Kular hospital, Punjab, India. Patients who underwent tailored MGB-OT between June 2008 and December 2009 were included. Primary outcomes of interest included a variety of weight loss outcome measures including % Excess Weight Loss (%EWL) at 1, 5 and 10 years in relation to a "tailored" Bilio-Pancreatic Limb Length (BPLL.)

The study was motivated by questions raised suggesting that a BPLL in the OAGB (MGB-OT) should be limited to 150 cm. Data were collected with a team of nurses and support staff that maintained a daily calling and follow up list adding data to an easily accessible online electronic database.

The analytic process assessed various weight loss outcomes at 1, 5 and 10 years following "tailored" BPLLs in patients undergoing the Mini-Gastric Bypass Original Technique (MGB-OT) as described by Rutledge. In addition to using simple statistical methods to assess the relation of the BPLLs to weight loss outcomes, a linear regression model was used to analyse and quantify the relationship between the length of the tailored BP limb and the weight loss measures a 1, 5 and 10 years after operation.

The study design focused upon the "power" of the BPLL as measured by 1, 5 and 10 year weight loss outcomes. The study was designed to answer two specific questions: first is a "FIXED" BPLL of 150 cm best for everyone (I.e. like the fixed BPLL used in the RNY) or put differently: is a 150 cm BPLL equally efficacious as compared to a longer BPLL when judged by measures of weight loss at 1, 5 and 10 years after surgery. Analysis included comparing BPLLs to the various 1, 5 and 10 year weight loss measures such as BMI, %BMI lost, Total weight at 10 years, % Excess Weight Loss at 10 yrs and other standard outcome measures.

Further, if such a relationship does indeed exist, can it be more precisely quantified? For example, is it "linear," that is to say for each and every additional cm of BPLL do the various long term weight loss measures increase similarly?.

There are of course many other questions now in bariatric surgery and related to the MGB/OAGB but the present study was designed to be sharply focused upon these two questions. Risk benefit and predictive power and multivariate analysis and creation of guidelines are in process and have been addressed in the past and will be part of subsequent publications., , ,

Notably the government of India health-care system provides no support for bariatric surgery and specifically no support at all for the MGB at any time during the course of this study and up until the time of this writing. All patients in the study paid out of pocket for the operation. The self pay situation and the fact that poor outcomes are little tolerated are also worthwhile noting. Given this climate and the capped hospital resources in a small town, it has been remarkable that the surgeons in this study have maintained a sterling record of excellent outcomes, a busy clinical practice with outcomes and results that rival those reported from other areas of the world including some of the best hospitals in the United States. The "tailored" MGB-OT used by the surgeon authors facilitated excellent outcomes and supported their success even in such demanding circumstances.

Once a significant association between BPLL and outcomes was determined, then a linear regression analysis was performed to further quantitate and describe the relationship between BPLL and outcome measures.

The present small first step is part of a longer term effort to investigate creation of a tool so robust that it might act as a guide for both patients and surgeons who might select the MGB-OT.

The study was conducted in accordance with the principles of the Declaration of Helsinki. Ethical permission was obtained from the local ethics committee and all participants provided written informed consent for data sharing.

ELIGIBILITY:
Inclusion Criteria: Patients selected for Mini-Gastric Bypass - Original Technique at Kular Hospital -

Exclusion Criteria: None

-

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients selected for Mini-Gastric Bypass - Original Technique at Kular Hospital
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Percent Excess Weight Loss | 10 years following operation
  Amount of weight lost assessed by Percent Excess Weight Loss
Percent Total Weight Loss | 10 years following operation
  Amount of weight lost assessed by Percent of Total Weight Loss

CONTACTS AND LOCATIONS:
Overall Officials: R Rutledge, MD, Principal Investigator — Kular Hospital
Locations (1):
- Kular Hospital, Khanna, Punjab, India

IPD SHARING:
Plan to Share IPD: No